CLINICAL TRIAL: NCT05984836
Title: Safety Starts at Home: Nursing Led Education Toward Enhancing Mothers' Knowledge and Attitude Regarding Early Childhood Injuries.
Brief Title: Early Childhood, Home Injuries, Mothers ' Knowledge, Mothers' Attitude
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Matrouh University (Other)
Responsible Party: Principal Investigator, Seham El-Sayed Saleh Hassan, Lecturer of pediatric nursing, faculty of nursing, Matrouh University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: IRB00013620(9/19/2025)
Record Dates: First submitted 2023-07-12; First posted 2023-08-09 (Actual); Last update posted 2025-04-02 (Actual); Status verified 2025-03

CONDITIONS: Home Injury
Keywords: Home injuries; Early childhood; Rural mothers; First aid

STUDY DESIGN:
Intervention Model Description: Find out the impact of Early Childhood Home-Related Injuries education on the Mothers' Knowledge and Attitudes regarding First Aid in Matrouh.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- health education class (Experimental): Those mothers receive Early Childhood Home-Related Injuries education regarding First Aid in Matrouh
  Interventions: Behavioral: Implement health education
- Control group (No Intervention): Those mothers not receive Early Childhood Home-Related Injuries education regarding First Aid in Matrouh

INTERVENTIONS:
Behavioral: Implement health education — Implement health education class for the rural mothers in the for of one session will take about 30 minutes and it will include the following:
  First aid (fracture, burn, bleeding, injuries and food poising). Critique malpractice for injuries management behavior at home.
  About 10 mothers will be included in the session. Each session will take 30 minutes (in the family health center), to cover all theoretical contents.
  The researcher will use different teaching methods as demonstration and discussion, learning aids as handout, video and pictures.
  Arms: health education class

SUMMARY:
Home-Related Injuries among Early Childhood: Rural Mothers' Knowledge, Attitudes and Practice regarding First Aid in Matrouh Governorate, Egypt

Keywords: Home injuries, Early childhood, Rural mothers, First aid, Matrouh Governorate.

DETAILED DESCRIPTION:
Implement health education class to rural mothers about first aid measures to be taken for their injured children"

ELIGIBILITY:
Inclusion Criteria:

* The Mothers have normal preschool children less than 6 years regardless the child gender.
* Educated (minimum accepted level of education is completion of primary education)
* Interested & willing to participate in the study.

Exclusion Criteria:

-

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Mothers of children under five years
Enrollment: 400 (Actual)
Dates: Start 2023-05-25 (Actual); Primary Completion 2023-12-30 (Actual); Study Completion 2023-12-30 (Actual)

PRIMARY OUTCOMES:
Mothers' knowledge related First Aid Record | one session will take about 30 minutes
  This tool will be developed by the researcher after reviewing relevant literature to collect the required data from the mothers regarding first aid at home.
  It was developed by Bayomi and Mobarak (2013), translated to the Arabic language to assess mothers' knowledge about home accidents in children. It consisted of 6 questions. Each question was given a score of zero or one. Correct answer questions had a score of one and incorrect answers had a score of zero. Total score was classified as poor knowledge (<50%), moderate knowledge (50%-75%), and good knowledge (>75%).
  * Part (3): 25-item questions to assess the practice and attitude of mothers towards home-related injuries. Eight negative and 17 positive items were developed (Likert scale rate).
  * Part 4: Mother's Subjective Practices regarding to first aid at home scale. This part will be developed by the researcher based on related literature (Network, 2009), (Fatouh et al., 2020), (KUMAR, SIDHU, & ZABI, 2020).

SECONDARY OUTCOMES:
Tool II: Mothers' Attitude related First Aid Record | 30 minutes
  This scale developed by Yalaki et al., )2010 (is a questionnaire aiming to identify attitudes of families towards home accidents. This tool was developed by (, translated to the Arabic language to measures mothers' attitude toward first aid. It consists of 25 questions to assess mothers' attitudes and practice toward first aid. Eight negative and 17 positive items were developed (Likert scale ratio). Responses: "always -frequently" and "sometimes-rarely-never" were measured together.
  Positive answers question were scored as one point, while negative answers were scored as a zero point. The total score was categorized as negative attitude [zero to 12 (< 50%)], neutral attitude [13-18 (50% -75%)], and positive attitude [19-25 (> 75%)].

CONTACTS AND LOCATIONS:
Overall Officials: Seham Saleh, Lecturer, Principal Investigator — Matrouh University
Locations (1):
- Matrouh university, Marsá Maţrūḩ, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Al-Bshri SA, Jahan S. Prevalence of home related injuries among children under 5 years old and practice of mothers toward first aid in Buraidah, Qassim. J Family Med Prim Care. 2021 Mar;10(3):1234-1240. doi: 10.4103/jfmpc.jfmpc_2265_20. Epub 2021 Apr 8. PMID 34041157
- [Background] Anwar M, Mostafa Z, Elareed H. Maternal Knowledge and Attitude about Home-related Injuries in Children under the Age of Five Years. Egyptian Family Medicine Journal (EFMJ) 2021; 5(2). 1-105. http://efmj.journals.ekb.eg/
- [Background] Bagahirwa I, Mukeshimana M, Cherian T, Nkurunziza T, El-Khatib Z, Byiringiro JC, Ng'ang'a L, Rusingiza E, Riviello R, Ndayisaba GF, Hedt-Gauthier BL. Presentation of Pediatric Unintentional Injuries at Rural Hospitals in Rwanda: A Retrospective Study. Ann Glob Health. 2020 Sep 14;86(1):116. doi: 10.5334/aogh.2711. PMID 32983912
- [Background] Centers for Disease Control and Prevention, National Center for Injury Prevention and control. Injuries Among Children and Teens.2021. https://www.cdc.gov/injury/features/child-injury/index.html#Child-Injury-Deaths-Data
- [Background] Eldosoky RS. Home-related injuries among children: knowledge, attitudes and practice about first aid among rural mothers. East Mediterr Health J. 2012 Oct;18(10):1021-7. doi: 10.26719/2012.18.10.1021. PMID 23301356
- [Background] Mohammed H, Wassif, Hakim S, Moustafa M. Frequency of Unintentional Home Injuries in Children under Five Years and its Relation with Environmental Risk Factors, Cairo, Egypt. The Egyptian Journal of Community Medicine, 2019; 37 (3). 93-102.
- [Background] Megahed M., Khalil N., Ibrahemc R., El Disoki R. Knowledge, attitude and practice of rural mothers towards home injuries among children under 5 years of age in Menoufia District- Menoufia Governorate, Egypt. Menoufia Medical Journal, 2016; 29 (4):1033-1039. DOI: 10.4103/1110-2098.202506
- [Background] Olutayo OG. Mother's Education, Age and Knowledge about Home Accident Prevention among Preschool Children in Ilesa Metropolitan City: A Relational Approach. Journal of Education and Practice, 2013; 4(11). 221-28
- [Background] Stephenson J. Caring for the injured child in settings of limited resource. Semin Pediatr Surg. 2016 Feb;25(1):19-22. doi: 10.1053/j.sempedsurg.2015.09.005. Epub 2015 Sep 16. PMID 26831134